CLINICAL TRIAL: NCT02347644
Title: Pilot Study of Prevention of Alcohol and Other Drug Use Using Motivational Interviewing Among Youth in Ukraine
Brief Title: Prevention of Substance Use in Youth in Ukraine
Acronym: PSUUKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Medical University, Ukraine (Other)
Responsible Party: Principal Investigator, Maureen A Walton, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D43TW009310 (NIH)
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Motivational Interview (Experimental): Given a brief motivational interview encouraging reduced use of alcohol and drugs.
  Interventions: Behavioral: Brief Motivational Interview
- Youth Control Group (No Intervention): Given a brochure with all available organizations in the community for help with alcohol and drug problems.

INTERVENTIONS:
Behavioral: Brief Motivational Interview — Motivational interviewing is a technique which aims to be both non-judgmental and non-confrontational. Its success depends largely on the presentation of objective feedback based on information provided by an individual. The technique involves acknowledgement that individuals who attend a counselling session, assessment or prevention program may be at different levels of readiness to change their alcohol consumption patterns, including:
  * No perception of any alcohol consumption problem
  * Realization of alcohol consumption problem with no corresponding action
  Arms: Brief Motivational Interview

SUMMARY:
The objective of this study is to explore the efficacy of brief motivational interventions (BMIs) for treatment of youth with alcohol and other drug problems after at least 3 months. The results of previous studies indicate that brief interventions for unhealthy alcohol use have been shown to be effective in primary care settings, with most studies focusing on adults and few studies focusing on youth. To date, no BMI studies have been conducted in the Ukraine among youth with alcohol or other drug use. Of particular concern are emerging adults ages 18-25 who may be at particularly high risk for alcohol problems given historical events related to the fall of the Soviet Union and the subsequent economic down turn.

This study will evaluate the efficacy of BMI by comparing BMI and no BMI conditions among two samples of youth screening positive on the prescreen survey for risky drinking. The subject pool will come from the Psychoneurological Department: the first location is located in the Railway Clinical Hospital, its clinical base, and the second in classes in the department at Kiev National Medical University.

The total sample of 120 will be broken down to 1.) 60 patients from Railway Clinical Hospital; and 2.) 60 students from Kiev National Medical University. Participants will be stratified by recruitment site and randomized to condition: BMI and control, with follow-up assessment at 3 months. In addition to being the first of study to evaluate the efficacy of BMI on substance use problems among youth in Ukraine, this study will examine BMI intervention processes in relation to alcohol and other drug outcomes. Findings will inform research and clinical practice to enhance early identification and prevention of problematic alcohol use trajectories among emerging adults

DETAILED DESCRIPTION:
Research Hypothesis

1. The rates and correlates of alcohol and other drug use, abuse and dependence, among young adults age 18-25 presenting to a Psychoneurological Department in the Railway Clinic Hospital in Kiev and Kyiv National Medical University will be high on the prescreen survey and may not be related to self-identification of problems.
2. The quality of life of young people with alcohol and substance use problems can be low compare to people without these problems. The quality of life can be improved after Brief Motivational Interventions.
3. The rates of intentional and unintentional injury (e.g., motor vehicle, violence related (fighting), sports injury, and other non-suicidal self-injury behavior) will be higher among emerging adults with greater alcohol and other drug use.
4. The Brief Motivational Interventions will help young people with alcohol and substance use problems and will be more effective for those with drinking motives that are social enhancement/externalizing and for those with less depression, anxiety levels, sleep disorders, impulsivity, sensation seeking, and aggression.
5. The Brief Motivational Interventions will help young people with alcohol and substance use problems and will found to be effective in reducing primary outcomes (alcohol and other drug use, as well as substance use related consequences) and secondary outcomes (depression and anxiety levels, sleep disorders, aggression, and quality of life).

Background According to the World Health Organization (WHO), youth in the Ukraine have the greatest level of alcohol consumption in the world, with typical age of initiation being 10 - 13 years old. When examining poisoning among youth in the Ukraine, 60% is caused by alcohol 3. Although the legal drinking age in the Ukraine is 18 for wine and liquor, beer is not legally classified as an alcoholic beverage and thus has no minimum drinking age. In 2011WHO ranked the Ukraine as 5th in the world in capita alcohol consumption. Recently, attempts have been made to address these issues. For example, in 2010 legislation was passed restricting access to low alcohol content beverages (e.g., beer) to youth, prohibiting access in various settings (i.e., public transportation, education, playgrounds, etc.).

Young adults are a particularly interesting cohort to examine in Ukraine, as these youth were raised following the downfall of the Soviet Union in 1991, during a socio-economic downturn. For example, data from the Ukrainian Longitudinal Monitoring Survey shows about 4 in 10 males and 1 in 10 females drank alcohol in the last month. Despite these alarming statistics, a paucity of data exists which examines correlates of alcohol use among young adults in Ukraine. Consistent with problem behavior theory, a variety of studies from the U.S. and Europe show that alcohol use and other problem behaviors tend to cluster during adolescence and young adulthood, likely due to shared risk and protective factors, with some researchers and clinicians viewing alcohol misuse as a self-harm behavior. Although commonly, self-harm has the connotation of an intentional, self-inflicted, physical injury or suicide attempt, substance use and eating disorders may be also considered non-suicidal self-harm behavior. Further, some researchers assign the choice of involvement with HRO (e.g., increased risk of injury including unintentional death) and the non-observance of safety rules during work as self-harm behaviors. The boundaries between suicide and non-suicidal self-harm behaviors are not always clearly defined, and in some cases behaviors that usually fall outside the boundaries of self-harm may indeed represent self-harm if performed with explicit intent to cause tissue damage. Self-harm is listed in the DSM-IV-TR as a symptom of borderline personality disorder or it can be a comorbid disorder. The motivations for self-harm vary, as it may be used to fulfill a number of different functions. For example, it may function as a coping mechanism, which provides temporary relief of intense feelings (e.g., anxiety, depression, stress, and emotional numbness), a sense of failure or self-loathing, or other mental traits including low self-esteem. Self-harm is most common during adolescence and young adulthood, usually first appearing between the ages of 12 and 24.

Early intervention for emerging adults with risky drinking may be a more effective use of resources than exclusive focus on treatment of those with alcohol use disorders (Nathan, 1988). A pilot study conducted in Ukraine survey emerging adults in an inpatient hospital and found that most did not think they had an alcohol problem. Further, our data found that common motives for alcohol use were related to coping with negative affect (e.g., stress, anxiety) and social influences (e.g., because my friends use alcohol). These findings are similar to that of American studies with college students, in which common motives for drinking included: coping-anxiety, coping-depression, social, enhancement, and conformity (Grant et al., 2007). In this regard, brief motivational interventions (BMIs) may be useful to enhance desire to change behavior and address motives for use in order to reduce risk of future alcohol problems. The need for early intervention may be particularly important for young adults with alcohol use and co-morbid anxiety and/or depression.

In spite of the available literature data about the problem of alcohol consumption there is the lack of information about efficacy of BMIs to reduce alcohol and other substance use among emerging adults in Ukraine. Among emerging adults in the U.S., studies suggest BMI approaches are promising among emerging adults.

In Europe, studies also showed the high efficacy of BMI in youth and adults. The goal of a German study was to gain knowledge about the target group of medically referred alcohol intoxicated adolescents and young adults, and to identify the utility of the administered BMI. Namely, researchers tried to find out more about the age and gender structure of participants, their alcohol and drug use history and their history of previous incidents of acute alcohol intoxication, their risky substance use and symptoms of psychopathology. Also, they assessed how many participants of the BMI took advantage of recommended further counseling regarding their alcohol use. Third, it was examined in what characteristics the group of "help accepters" differs from the group of "help avoiders" with regard to socio-demographic characteristics and substance use patterns. Yet, this research faced several limitations. First, the BMI was only semi-structured. It was uncontrolled stage- 1-design (there was not a control group); thus, researchers were not able to demonstrate the efficacy of the BMI. It remains unclear, if the BMI initiated change motivation or had the effect of motivational enhancement. The efficacy of the subsequent youth-specific counseling services was not examined. Another European study illuminates the existing evidence concerning the efficacy of brief motivational intervention [20]. Thus, there remain unanswered questions around the effectiveness of brief alcohol intervention across different settings, different population groups including emerging adults, about the optimal intervention content, and the longevity of intervention effects.

In this regard, a recent U.S. study in primary care used the Composite International Diagnostic Interview Alcohol Module to identify adults with alcohol problems in 3 randomized controlled trials comparing BMI with no BMI. These were conducted in the USA in order to identify key intervention components. This study examined 3 sets of audio-recorded BMIs (2 from null studies - no difference in drinking between BMI and no BMI groups; and 1 from a positive study - less drinking in BMI group compared with no BMI group). The drinking decreased among participants in all 3 studies. Intervention characteristics that are considered as central to efficacious BMIs (such as changes in self- or other reports of drinking quantity and/or frequency, drinking intensity and drinking within recommended limits) were not strong predictors of drinking outcome. The quality of the BMI processes was not predictive in these studies and may require attention to factors beyond constructs typically examined. Therefore, more detailed analysis and prospective studies are necessary. For example, the varying efficacy of BMI may depend on different factors such as drinking motives, impulsivity, depression, anxiety, sleep disorders, and aggression.

Study Design Over a one year period, this Psychoneurological Department based study will use a randomized controlled trial (RCT) design. Also, the Psychological Faculty of Kyiv National Medical University. Eligible young adults will complete a screening survey. Given the fact that we plan to include patients and students, we chose this subject pool for the study because it combines the psychiatric ward and base of students at the university. Those with risky drinking will be enrolled in the RCT and randomized to conditions and stratified by patient/student and given either the brief motivational intervention or the control brochure. A follow-up assessment will be conducted at 3 months.

Statistical Design

SPSS software version 18 will be used for data analysis. A regression model will be applied according to the distribution of the data.

ELIGIBILITY:
Inclusion Criteria:Adults ages 18-25 able to provide informed consent: 1) adults presenting to the Railway Clinic Hospital for a medical problems except for exclusion criteria below and, 2) students of KNMU ages 18-25. Additional inclusion criteria for the RCT is:

* have prescreen survey results indicating alcohol and drug abuse risk or have diagnosis of alcohol or substance use dependence according to ICD-10
* Between the ages of 18-25
* speaks and writes Ukrainian or Russian
* provide informed consent to participate

Exclusion Criteria: 1) Adults classified as "psychotic patients" (who need special treatment and are not able to follow the requirements of the protocol); (2) adults deemed unable to provide informed consent by hospital personnel or research staff (e.g., intoxication, mental incompetence) and (3) adults with suicide attempts in their history or with suicidal thoughts in the past (because they present in high psychological distress requiring intensive attention and intervention by staff); When we ask our patients about suicidal thoughts and acts, and we will evaluate the suicidal risk for clinical referral and because it is an important inclusion criteria. the patient has a high suicidal risk, If we see that a participant has suicidal thoughts, suicidal attempts or suicidal risk according to the results of the scales, we will we will exclude him/her from the study; provide medical care, and phone numbers and addresses of help desk, but will not take financial responsibility for that care. 4.) We will also exclude pregnant women.

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption at Time Two of Follow-up Survey | Three Months
  AUDIT-C total score, Q X F, Abstinence as defined as a day without any alcohol or drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, MPH, PhD, Principal Investigator — University of Michigan
Locations (2):
- University of Michigan Health System, Ann Arbor, Michigan, United States
- Kyiv National Medical University, Kyiv, Ukraine